CLINICAL TRIAL: NCT06288178
Title: The Effect of Consumption of Bread Types Made From Various Flours on Blood Glucose Fluctuations in Individuals With Obesity and Normal-Weight: A Randomized Controlled Trial
Brief Title: The Effect of Consumption of Bread Types Made From Various Flours on Blood Glucose Fluctuations
Acronym: Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Fatih Cesur, Assistant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/18
Record Dates: First submitted 2024-02-17; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Glycemic Index; Blood Glucose; Bread
Keywords: obesity; Glycemic index; Blood glucose; Cornbread; Buckwheat bread
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Types of bread (Experimental): The three breads (whole wheat bread, buckwheat bread, and cornmeal bread) contained 30 grams of digestible carbohydrates. Participants consumed these breads when they were hungry. Blood glucose was measured with a glucometer at 0 (fasting), 30, 60, 90, and 120 minutes. Anthropometric measurements were measured by BIA method and weight classification (obesity and normal weight) was made.
  Interventions: Dietary Supplement: Bread consumption
- Reference bread (White bread) (Experimental): Control group. Blood glucose comparison of all breads was determined according to white bread. The measurement method used was the same as for the other breads.
  Interventions: Dietary Supplement: Bread consumption

INTERVENTIONS:
Dietary Supplement: Bread consumption — There were four groups: whole wheat (WWB), buckwheat (BWB), corn bread (CB) and reference bread.

SUMMARY:
The obesities were aimed at the effect of whole wheat (WWB), buckwheat (BWB), and cornbread (CB) on blood glucose by comparing the glycemic index values with reference bread (RB).

Overall, WWB consumption had a positive effect on blood glucose in individuals with obesity, while BWB consumption caused an increase in blood glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* The study group consisted of volunteer individuals aged between 18 and 35 years.
* The first blood glucose measurement was taken after at least 8 hours of fasting and any of the bread types were given to the participants for consumption.
* All measurements were taken between 09.00-13.00.
* During the measurements, the volunteers were observed to avoid water, coffee, and any food intake and to avoid excessive exercise.

Exclusion Criteria:

* Pregnant,
* lactating women
* patients with physician-diagnosed chronic diseases
* Medication use

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
One loaf of bread was been consumed every week. Blood glucose measurements were performed with a glucometer at 0 (fasting), 30, 60, 90, and 120 minutes after each bread consumption. | Within research completion, an average of 4 week
  The effect of loaves of bread with a high glycemic index on blood sugar is well known. The higher the glycemic index, the higher the blood sugar fluctuation. Glycemic index values should be lower than white bread.

SECONDARY OUTCOMES:
This classification as obese and normal-weight individuals was made with the BIA (Bioelectrical impedance analysis) method. This classification was understood by anthropometric measurements made in the first week. | Within research completion, an average of 1 week
  It is known that high glycemic index values of bread consumption are paralleled by high blood fluctuations. On the other hand, the impact of bread consumption on obesity and normal weight people is also of interest. In obese people, the high glycemic index predisposes them to overeating. It can be said that the consumption of whole wheat bread caused lower blood glucose fluctuations than white bread, and on top of that, corn bread caused lower changes in blood glucose fluctuations than other breads in obese individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Avrasya University, Trabzon, Turkey (Türkiye)